CLINICAL TRIAL: NCT00005808
Title: Phase I Study Photodynamic Therapy Using Lutrin (Lutetium Texaphyrin) in the Treatment of Patients With Cervical Intraepithelial Neoplasia
Brief Title: Photodynamic Therapy Using Lutetium Texaphyrin in Treating Patients With Cervical Intraepithelial Neoplasia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively complete.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2012-02328; MWH-99-077; U01CA099168 (NIH); CDR0000067801 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia Grade 2; Cervical Intraepithelial Neoplasia Grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — motexafin lutetium; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

ARMS (2):
- Part 1 (lutetium texaphyrin, LEEP) (Experimental): Patients receive lutetium texaphyrin IV over 5-20 minutes. Patients undergo in vivo tissue assessment by spectrometer at 0, 1, 3, 5, 12, and 24 hours and loop electrical excision procedure (LEEP) at 24 hours after lutetium texaphyrin infusion.
  Interventions: Drug: motexafin lutetium; Procedure: loop electrosurgical excision procedure; Other: laboratory biomarker analysis
- Part 2 (lutetium texaphyrin, laser therapy, LEEP) (Experimental): Patients receive lutetium texaphyrin IV over 5-20 minutes. A laser delivers 730 nm of light to the cervix for 4, 8, or 16 minutes. Patients undergo LEEP at 4, 8, or 12 hours after exposure of the cervix to the light source.
  Interventions: Drug: motexafin lutetium; Drug: photodynamic therapy; Procedure: loop electrosurgical excision procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: motexafin lutetium — Given IV
  Other Names: Antrin; lutetium texaphrin; lutetium texaphyrin; Lutex; PCI-0123
Drug: photodynamic therapy — Undergo laser therapy
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
  Arms: Part 2 (lutetium texaphyrin, laser therapy, LEEP)
Procedure: loop electrosurgical excision procedure — Undergo LEEP
  Other Names: LEEP; Loop Electrosurgical Excision
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the effectiveness of photodynamic therapy with lutetium texaphyrin in treating patients who have cervical intraepithelial neoplasia. Photodynamic therapy uses light and drugs such as lutetium texaphyrin that make abnormal cells more sensitive to light and may kill abnormal cells in the cervix and prevent the development of cervical cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the optimal dosage with the least toxicity of lutetium texaphyrin as well as the length of time following its systemic injection that provides the maximum differential in drug uptake between the target dysplastic squamous cells and normal squamous epithelium when given to patients with cervical intraepithelial neoplasia (CIN).

II. Determine, by histomorphometry, the photodynamic light dose that demonstrates the greatest treatment selectivity between normal cervical epithelium and CIN with the least amount of cervical pain and necrosis.

OUTLINE: This is a dose-escalation study of lutetium texaphyrin (part 1) followed by a dose-escalation study of light fluence (part 2).

Part 1: Patients receive lutetium texaphyrin IV over 5-20 minutes. Patients undergo in vivo tissue assessment by spectrometer at 0, 1, 3, 5, 12, and 24 hours and loop electrical excision procedure (LEEP) at 24 hours after lutetium texaphyrin infusion.

Part 2: Patients receive lutetium texaphyrin IV over 5-20 minutes. A laser delivers 730 nm of light to the cervix for 4, 8, or 16 minutes. Patients undergo LEEP at 4, 8, or 12 hours after exposure of the cervix to the light source.

Cohorts of 9 patients receive escalating doses of lutetium texaphyrin (part 1) and then light fluence (part 2) until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which 2 of 9 patients experience dose-limiting toxicity.

Patients are followed at 48 hours, weekly for 1 month, and then at 4 months.

PROJECTED ACCRUAL: A maximum of 54 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Cervical intraepithelial neoplasia (CIN) grade II or III
* No cytologic, colposcopic, or histologic evidence of invasive squamous cell carcinoma
* No evidence of glandular atypia on Pap smear, endocervical curettage, or biopsy
* No inadequate colposcopy (i.e., entire transformation zone cannot be visualized and/or upper limit of a colposcopically abnormal lesion cannot be visualized fully)
* HIV positive but not currently on antiviral therapy
* Performance status - 0-2
* WBC greater than 4,000/mm^3
* Absolute neutrophil count greater than 2,000/mm^3
* Platelet count normal
* Liver enzymes normal
* No liver impairment
* BUN normal
* Creatinine normal
* No renal insufficiency
* No coronary artery disease
* No cardiac arrhythmia
* No congestive heart failure
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for at least 1 month after study
* No other serious medical illness (e.g., non-insulin and insulin-dependent diabetes or connective tissue disorders)
* No other prior or concurrent malignancy
* No known G6PD deficiency
* No porphyria
* No history of 2 prior ablative/excisional therapies (i.e., cryotherapy, laser ablation, loop electrical excision procedure, or cold knife cone biopsy)
* No concurrent non-steroidal anti-inflammatory drugs (NSAIDS)
* No other concurrent significant medication/therapy such as:
* Anti-hypertensives, anti-arrhythmics, or inotropic agents for cardiopulmonary disease
* Diuretics for renal insufficiency
* Steroids or NSAIDs for connective tissue disorders

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2000-12; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Optimal dosage with the least toxicity of lutetium texaphyrin (Part 1) | Up to 24 hours
  A simplified graphical analysis will be utilized to determine the drug dose and time after administration that provides the largest differential area between lutein texaphyrin tissue levels in neoplastic and normal cervical tissue
Maximal differential in Lutrin tissue levels between normal and dysplastic cells (Part 1) | At the time of LEEP
Percentage of tissue demonstrating PDT related effects (apoptosis/ necrosis) for normal versus abnormal epithelium at each total fluence for each LEEP cone biopsy specimen | At LEEP time
  A simplified graphical analysis will be utilized to determine the fluence that provides the maximal differential area between neoplastic and normal cervical epithelium and stroma.

CONTACTS AND LOCATIONS:
Overall Officials: John Comerci, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States